CLINICAL TRIAL: NCT00007475
Title: Permeability Factor in Focal Segmental Glomerulosclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010053; 01-DK-0053 (Other: National Institutes of Health)
Record Dates: First submitted 2000-12-22; First posted 2000-12-25 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: Plasma Exchange; Cyclophosphamide; Proteinuria; Hemodialysis; Expression Profiling
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria | interventions — Plasma Exchange; Plasmapheresis; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plasma Exchange + Cyclophosphamide (Experimental): Procedure/Surgery: Plasma exchange A course of plasma exchange of 5 treatments over 10 days, then administration of cyclophosphamide.
  Drug: Cyclophosphamide For GFR > 50 ml/min/1.73 m2 received oral cyclophosphamide at a dose of 2 mg/kg/ day for 3 months. For GFR < 50 ml/min/1.73 m2 but > 10 ml/min/1.73 m2 will receive oral cyclophosphamide at a 25% reduced dose or 1.5 mg/kg/d for 3 months.
  Interventions: Procedure: Plasma exchange; Drug: Cyclophosphamide

INTERVENTIONS:
Procedure: Plasma exchange — A course of plasma exchange of 5 treatments over 10 days, then administration of cyclophosphamide.
  Other Names: Plasmapheresis
Drug: Cyclophosphamide — For GFR > 50 ml/min/1.73 m2 received oral cyclophosphamide at a dose of 2 mg/kg/ day for 3 months. For GFR < 50 ml/min/1.73 m2 but > 10 ml/min/1.73 m2 will receive oral cyclophosphamide at a 25% reduced dose or 1.5 mg/kg/d for 3 months.
  Other Names: Cytophosphane

SUMMARY:
Focal segmental glomerulosclerosis (FSGS) is a renal syndrome characterized by proteinuria (usually nephrotic range), limited response to conventional therapy, and a poor renal prognosis, with progression to end stage renal failure in at least 50% of patients. As a syndrome, FSGS likely has many specific etiologies, only a few of which are well-defined. Recently, it has been suggested that some idiopathic FSGS patients have elevated circulating levels of a protein that induces glomerular permeability in vitro and in vivo. While there has been no consistent term for this factor, it will be termed here FSGS permeability factor (FPF).

The purposes of the present study are five fold:

1. To identify a population of FSGS patients with elevated FPF levels
2. To examine RNA expression profiles of peripheral blood mononuclear cells (PBMC) in FSGS patients with elevated FPF levels
3. To define the kinetics of FPF disappearance and reappearance in FSGS patients receiving immunomodulatory therapy and in the case of patients with recurrent FSGS following renal transplant, those receiving plasma exchange
4. To identify immunosuppressive agents which are successful in inducing sustained reduction in FPF levels
5. To determine in patients with FSGS who are awaiting renal transplant, whether sustained reduction in FPF levels is associated with reduced risk of recurrent FSGS.

Patient participation is divided into an evaluation phase, in which FPF levels, RNA expression profiles, and patient eligibility for participation in treatment protocols are determined, and a treatment phase in which specific immunomodulatory therapy is introduced in an open label fashion. We propose to define carefully the relationship between elevated FPF and remission of proteinuria in patients with FSGS in native kidneys, following treatment with standard therapies (daily prednisone, cyclophosphamide) and experimental therapies (pulse dexamethasone, pirfenidone). In patients with recurrent FSGS in renal allografts, we will determine the kinetics of FPF following plasma exchange and following plasma exchange plus cyclophosphamide. In patients with elevated FPF levels who are awaiting renal transplantation, we will determine the kinetics of FPF following plasma exchange and following plasma exchange plus cyclophosphamide, and examine the rate of recurrent FSGS in these patients.

DETAILED DESCRIPTION:
Focal segmental glomerulosclerosis (FSGS) is a renal syndrome characterized by proteinuria (usually nephrotic range), limited response to conventional therapy, and a poor renal prognosis, with progression to end stage renal failure in at least 50% of patients. As a syndrome, FSGS likely has many specific etiologies, only a few of which are well-defined. Recently, it has been suggested that some idiopathic FSGS patients have elevated circulating levels of a protein that induces glomerular permeability in vitro and in vivo. While there has been no consistent term for this factor, it will be termed here FSGS permeability factor (FPF).

The purposes of the present study are five fold:

1. To identify a population of FSGS patients with elevated FPF levels
2. To examine RNA expression profiles of peripheral blood mononuclear cells (PBMC)

   in FSGS patients with elevated FPF levels
3. To define the kinetics of FPF disappearance and reappearance in FSGS patients

   receiving immunomodulatory therapy and in the case of patients with recurrent FSGS

   following renal transplant, those receiving plasma exchange
4. To identify immunosuppressive agents which are successful in inducing sustained

   reduction in FPF levels
5. To determine in patients with FSGS who are awaiting renal transplant, whether

sustained reduction in FPF levels is associated with reduced risk of recurrent FSGS.

Patient participation is divided into an evaluation phase, in which FPF levels, RNA expression profiles, and patient eligibility for participation in treatment protocols are determined, and a treatment phase in which specific immunomodulatory therapy is introduced in an open label fashion. We propose to define carefully the relationship between elevated FPF and remission of proteinuria in patients with FSGS in native kidneys, following treatment with standard therapies (daily prednisone, cyclophosphamide) and experimental therapies (pulse dexamethasone, pirfenidone). In patients with recurrent FSGS in renal allografts, we will determine the kinetics of FPF following plasma exchange and following plasma exchange plus cyclophosphamide. In patients with elevated FPF levels who are awaiting renal transplantation, we will determine the kinetics of FPF following plasma exchange and following plasma exchange plus cyclophosphamide, and examine the rate of recurrent FSGS in these

patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients with idiopathic focal segmental glomerulosclerosis on renal biopsy, including the following categories:

     A) Untreated FSGS

     B) Steroid-dependent FSGS

     C) Steroid resistant FSGS

     D) Recurrent FSGS, with functioning allograft

     E) FSGS in ESRD, receiving hemodialysis
  2. Adults greater than or equal to18 will be eligible for all studies.
  3. Children greater than 20 kilograms, will be eligible for all branches of the study except for treatment of steroid resistant FSGS with pirfenidone, as pirfenidone has not previously been administered to pediatric patients in any setting. Children less than 20 kilograms will be excluded from the study for the following reason: plasma exchange in patients less than 20 kilograms requires a red blood cell transfusion, which significantly increases the risk of the procedure by exposing the patient to the risk of transfusion associated infections, and the safety of an aggressive course of plasma exchange has not been established in this population.

EXCLUSION CRITERIA:

1. Secondary FSGS: HIV-associated FSGS or hyperfiltration FSGS, including FSGS associated with congenital renal abnormalities, renal mass reduction, reflux nephropathy, interstitial nephritis, and sickle cell anemia are excluded.
2. Patients with disease associated with immunosuppression, other than chronic renal failure.
3. The presence of malignancy or the history of other serious, complicating illness such as myocardial infarction or cerebrovascular accident in the past six months, at the discretion of the investigators.
4. For plasma exchange: A Department of Transfusion Medicine consultant will evaluate all potential plasma exchange patients. Those with prolonged PT, PTT, platelet count less than 100,000 or receiving anticoagulant therapy will undergo plasma exchange only if the consultant considers this to be safe.
5. For prednisone: uncontrolled diabetes mellitus (requiring greater than 100 units of insulin/day with the concurrence of the Endocrinology consultant), active infection including hepatitis B or C (if that is the advice of the Hepatology consultant), infection with HIV (as these patients are at increased risk of avascular necrosis), other active infection (if that is the advice of the Infectious Disease consultant), history of avascular necrosis or bone densitometry indicating bone mass less than 2SD below normal, active ulcer disease, history of steroid-induced psychosis, morbid obesity, positive PPD or history of past positive PPD without adequate treatment are excluded.
6. For Cyclophosphamide:

A) Allergy or hypersensitivity to cyclophosphamide

B) Leukocyte less than 3000 cells/microliter or ANC less than 1500 cells/microliter or evidence of bone marrow compromise

C) Prior irradiation to the heart or therapy with doxorubicin or other cardiotoxic medication (may increase the risk for cardiotoxicity)

D) Peritoneal dialysis, as there is no published evidence that cyclophosphamide metabolites can be safely removed.

E) Certain drugs will be used with caution or avoided. Barbiturates and phenytoin induce the hepatic enzymes that metabolize cyclophosphamide and therefore if these medications are required, cyclophosphamide doses may need to be increased to achieve a comparable immunosuppressive effect. Drugs that inhibit cyclophosphamide metabolism include allopurinol, imipramine, and phenothiazines, chloramphenicol and chlorpromazine; these drugs will be avoided. NSAID increase the risk of hyponatremia; these drugs will be avoided.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Kopp, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Korbet SM. Primary focal segmental glomerulosclerosis. J Am Soc Nephrol. 1998 Jul;9(7):1333-40. doi: 10.1681/ASN.V971333. No abstract available. PMID 9644647
- [Background] Cameron JS. Recurrent renal disease after renal transplantation. Curr Opin Nephrol Hypertens. 1994 Nov;3(6):602-7. doi: 10.1097/00041552-199411000-00007. PMID 7881983
- [Background] Valeri A, Barisoni L, Appel GB, Seigle R, D'Agati V. Idiopathic collapsing focal segmental glomerulosclerosis: a clinicopathologic study. Kidney Int. 1996 Nov;50(5):1734-46. doi: 10.1038/ki.1996.493. PMID 8914044

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment of subjects occurred at fraction of the anticipated rate despite over a decade of study conduct; the discrepancy between actual (15) and projected (100) enrollment is due to (a) lack of revising the registry entry with revisions of the protocol (n=50, excluding historical controls) and (b) lower referral rates by external nephrologists.
Groups:
- FPF NOT Assayed, Plasma Exchange + Cyclophosphamide Completed: Participants not assayed for FSGS Permeability Factor (FPF) levels pre-treatment (Tx), yet still complete both series of protocol-specified treatment; FPF levels NOT available as its assay has not yet been developed to an extent that it could be applied to all enrollees of this current trial
- FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed: Protocol Groups A/B/C (FPF < 0.6); group size is limited due to limited availability of provisionally validated FPF assay and discrepancy with protocol groups due to low-FPF participants receiving PE and Cyclophosphamide (contrast to protocol Figure 1)
- FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed: Protocol Group D (FPF 0.6 or greater pre-initial Transplant); group size is limited due to limited availability of provisionally validated FPF assay and discrepancy with protocol groups due to low-FPF participants receiving PE and Cyclophosphamide (contrast to protocol Figure 1)
- Historical Controls: Noted as Group F in study protocol: historical control patients, including patients at NIH or other institutions who have previously undergone renal transplant, for whom stored sera are available, and for whom consent to measure FPF has been can be obtained. In some cases, these measurements have been performed by Dr. Savin under pre-existing protocols and these data are already available.
Period: Overall Study
Arm/Group | FPF NOT Assayed, Plasma Exchange + Cyclophosphamide Completed | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed | Historical Controls
Started | 12 ([ arm reflects un-assayed participants' disposition ]) | 1 ([ arm reflects eventual participant disposition ]) | 2 ([ arm reflects eventual participant disposition ]) | 0
FSGS Permeability Factor (FPF) Assayed | 0 (FSGS Permeability Factor's provisional assay only applied to minority of early enrollees, by design.) | 1 | 2 | 0
Initial Transplant | 12 | 1 | 2 | 0
Post-initial Transplant Proteinuria | 12 | 1 | 2 | 0
Initial Plasma Exchange | 12 | 1 | 2 | 0
Initiate Cyclophosphamide | 12 | 1 | 2 | 0
Completed | 8 | 1 | 2 | 0
Not Completed | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FPF NOT Assayed Provisionally, PE + Cyclophosphamide Completed: Participants not provisionally assayed for FPF, yet still complete both series of protocol treatment: Plasma Exchange (PE) and Cyclophosphamide; note that these form a majority of enrollees due to limited availability of validated FPF assay (such an assay has not yet been developed to an extent that it could be applied to all enrollees of this current trial; see Outcome Measures for more details)
- FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed: Protocol Groups A/B/C (FPF < 0.6); group size is limited due to limited availability of validated FPF assay and discrepancy with protocol groups due to low-FPF participants receiving PE and Cyclophosphamide (contrast to protocol Figure 1)
- FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed: Protocol Group D (FPF 0.6 or greater pre-initial Transplant); group size is limited due to limited availability of validated FPF assay
- Total: Total of all reporting groups
Arm/Group | FPF NOT Assayed Provisionally, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed | Total
Number analyzed (Participants) | 12 | 1 | 2 | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years at consent] | 39.5 [32.25 to 47.25] | 63 [63 to 63] | 19 [18.5 to 19.5] | 37 [25 to 48.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 1 | 9
  Male | 4 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 6 | 1 | 2 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 1 | 2 | 15
Treated for Prior Recurrence [Number; unit: participants]
  Yes | 2 | 1 | 0 | 3
  No | 10 | 0 | 2 | 12
Time from onset/diagnosis of Focal Segmental Glomerulosclerosis to study enrollment/consent [Median (Inter-Quartile Range); unit: years] — Note: calculated in terms of whole years, subject to coarsening due to integer subtraction (whole-year age at consent - whole-year age at onset)
  years | 10 [7.75 to 14.75] | 6 [6 to 6] | 1.5 [1.25 to 1.75] | 8 [4 to 13.5]

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Proteinuria in Recurrent FSGS Following Renal Transplant With Plasma Exchange and Cyclophosphamide.
Description: Outcomes for FSGS occurring in native kidneys:
  A. Complete remission: proteinuria <0.3 g/d ; B. Partial remission: proteinuria between 0.3 and 2 g/d ; C. Incomplete response: proteinuria between 2 and 3.5 g/d ; D. Relapse: return to proteinuria ≥3.5 g/d ; Note that counts within each category A-D may be summarized relative to remaining categories, as a proportion (relative to complement of the whole group count) with calculations implicitly based on zero/one valued binary variables, whose means are proportions, so to report 95% confidence intervals calculated using an exact binomial distribution.
Time Frame: every 3 months up to a year followed with native kidneys
Population: all participants, regardless of amount of follow-up
Measure: Mean (95% Confidence Interval); unit: proportion of participants with outcome
Groups:
- FPF NOT Assayed, Plasma Exchange + Cyclophosphamide Completed: Participants complete both series of protocol treatment, Plasma Exchange and Cyclophosphamide.
- FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed: Protocol Group D (FPF 0.6 or greater pre-initial Transplant)
Arm/Group | FPF NOT Assayed, Plasma Exchange + Cyclophosphamide Completed | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed
Number analyzed (Participants) | 12 | 1 | 2
proportion of participants with outcome
  A. Complete remission: proteinuria <0.3 g/d | 0 [0 to 0.00049] | 0 [0 to 0.975] | 0.5 [0.01258 to 0.9874]
  B. Partial remission: proteinuria in [0.3,2] g/d | 0.25 [0.05486 to 0.5719] | 0 [0 to 0.975] | 0 [0 to 0.8419]
  C. Incomplete response: proteinuria in (2,3.5) g/d | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  D. Relapse: return to proteinuria ≥3.5 g/d | 0.1667 [0.02086 to 0.4841] | 1 [0.025 to 1] | 0 [0 to 0.8419]
Statistical Analysis 1: Comparison: FPF NOT Assayed, Plasma Exchange + Cyclophosphamide Completed vs FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed vs FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed; No groups compared, yet null hypothesis: pooled proportion = 0, tested using counts pooled across baseline FPF assay-availability groups (7 across 3 arms) excluding 4 non-completers (yielding 7/11 with event below). Given the modest group-specific sample sizes and tendency for zero outcomes to be observed in a group, we employ exact binomial 95% confidence intervals using the method of Clopper and Pearson (1934; calculated along with corresponding tests using Michael Fay's exactci package in R); Test type: Superiority or Other; p < 0.0001, Exact binomial test — Exact binomial test of proportion of participants exhibiting reduction in proteinuria (see definition below), under null hypothesis that the overall proportion is zero; Tested under null hypothesis that the overall proportion is zero; Proportion with reduced proteinuria = 0.6363, 95% CI 2-sided [0.3079 to 0.8907], Standard Error of Mean 0.0698 — Proportion event definition: exhibiting reduction in proteinuria post-cyclophosphamide (complete- [urine protein {UP} <0.3] or or partial-remission [between 0.3 & 2.0, inclusive], limited response [UP between 2.0 & 3.5] yet no relapse [UP 3.5+])

2. Secondary Outcome: Comparison of RNA Expression Profiles in PBMC From Patients With FPF, Without FPF and Control Subjects
Description: No RNA expression profiles have been obtained as FSGS Permeability Factor (FPF) levels NOT available -- its assay has not yet been developed to an extent that it could be applied to all enrollees of this current trial.
  Note that provisional values (targeting current candidate molecule: cardiotrophin-like cytokine 1) were assayed for 3 of the first 4 enrollees using assay by Dr. Virginia Savin, whose lab is actively investigating a molecular identification of FPF using an isolation approach based on sequential precipitation results in a 100-fold purification, but the fraction remains a complex mixture on SDS-PAGE (Sharma 1999). Other investigators of FPF include:
  1. Terry Phillips at NIH developed an assay that looked promising but after his retirement it has not been possible for other researchers to get this working.
  2. Avi Rosenberg, NCI has developed a promising ELISA-style assay, as well as some work in a mass spectrometry assay, and this is being further refined.
Time Frame: End of study
Population: Participants with FPF, without FPF and control subjects who have also had RNA expression profiling done in PBMCs.
Groups:
- FPF NOT Assayed, Plasma Exchange + Cyclophosphamide Completed: Participants complete both series of protocol treatment: Plasma Exchange + Cyclophosphamide
Arm/Group | FPF NOT Assayed, Plasma Exchange + Cyclophosphamide Completed | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Define the Kinetics of FPF in FSGS Patients Receiving Immunomodulatory Therapy or Plasma Exchange.
Description: Provisional assay of a molecular identification of FPF (current candidate: cardiotrophin-like cytokine 1) using an isolation approach based on sequential precipitation results in a 100-fold purification.
  Note: Focal segmental glomerulosclerosis Permeability Factor (FPF) assay had not yet been developed to an extent that it could be applied to all enrollees in the current trial; provisional values were assayed for 3 of the first 4 enrollees using a version implemented by Dr. Virginia Savin, whose lab is actively investigating the above isolation approach, but the fraction remains a complex mixture on SDS-PAGE (Sharma 1999). Other investigators of FPF, mentioned here for interested readers of this trial report, include:
  1. Terry Phillips at NIH developed an assay that looked promising prior to his retirement.
  2. Avi Rosenberg, NCI has developed promising ELISA-style assay, and mass spectrometry assay, being refined.
Time Frame: End of study
Measure: Mean (Full Range); unit: 1- albumin glomerular permeability ratio
Groups:
- Plasma Exchange + Cyclophosphamide, Complete Treatment: Participants complete both series of protocol treatment
Arm/Group | Plasma Exchange + Cyclophosphamide, Complete Treatment | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed
Number analyzed (Participants) | 0 | 1 | 2
1- albumin glomerular permeability ratio |  | 0.41 [0.41 to 0.41] | 0.865 [0.82 to 0.91]

4. Secondary Outcome: Correlate the Effect of Immunosuppressive Agents Which Reduce Proteinuria in Recurrent FSGS With the Effect on FPF Levels
Description: as for outcome 3
Time Frame: End of study
Population: Participants with FPF levels assayed following immunosuppressive therapies (currently none). Note: its assay had not yet been developed to an extent that it could be applied beyond the provisional values assayed for 3 of the first 4 enrollees using a version implemented by Dr.Virginia Savin, VA Medical Center/Kidney Institute, Kansas City, Missouri
Arm/Group | Plasma Exchange + Cyclophosphamide, Complete Treatment | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Determine Whether Renal Transplantation in Patients Whose Elevated FPF Levels Have Been Reduced for a Sustained Period is Associated With a Reduced Prevalence of Recurrent FSGS.
Description: as for outcome 3
Time Frame: End of study
Population: Participants whose post-transplantation follow-up yields 1 or more assayed FPF levels
Arm/Group | Plasma Exchange + Cyclophosphamide, Complete Treatment | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Entire course of study follow-up, from study enrollment to closure
Groups:
- Plasma Exchange + Cyclophosphamide, Complete Treatment: Participants for whom the Focal Segmental Glomerulosclerosis (FSGS) Permeability Factor, or FPF was not able to be assayed, yet enrolled and completed both protocol-specified interventions: the plasma exchange procedure and treatment by cyclophosphamide.
- FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed: Original protocol Groups A/B/C (FPF < 0.6); group size is limited due to limited availability of validated FPF assay and discrepancy with protocol groups due to low-FPF participants receiving PE and Cyclophosphamide (contrast to protocol Figure 1)
- FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed: Original protocol Group D (FPF 0.6 or greater pre-initial Transplant)
Arm/Group | Plasma Exchange + Cyclophosphamide, Complete Treatment | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/12 | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plasma Exchange + Cyclophosphamide, Complete Treatment (N=12) | FPF Assayed Pre-Tx as Low, PE + Cyclophosphamide Completed (N=1) | FPF Assayed Pre-Tx as High, PE + Cyclophosphamide Completed (N=2)
Rejection of Kidney Graft (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — Determined after 1 week of cyclophosphamide treatment
Hemorrhagic cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — BK viral infection confirmed by high urine BK count per mil 14 weeks after cyclophosphamide initiation; managed by NIH urology team
Adenocarcinoma of the Prostate Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — diagnosed at a point six weeks into treatment by cyclophosphamide
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — As defined in Protocol for Patient group 4 (Recurrent FSGS with functioning allograft), having a nadir ANC <500 cells/µl during cyclophosphamide treatment is a serious AE

LIMITATIONS AND CAVEATS:
Note: definitive FSGS Permeability Factor (FPF) assays still in development. Data/samples transferred to the NIH-CC Glomerulosclerosis Consolidation protocol: focus on cardiotrophin like cytokine 1 & antibodies to a panel of podocyte proteins as FPF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes